CLINICAL TRIAL: NCT03292562
Title: A Comparison of Methods of Discontinuing Nasal CPAP in Premature Infants <30 Weeks Gestation - a Feasibility Study
Brief Title: A Comparison of Methods of Discontinuing Nasal CPAP in Premature Infants <30 Weeks Gestation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Amir Mustafa Khan, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC-MS-17-0334
Record Dates: First submitted 2017-09-21; First posted 2017-09-25 (Actual); Results first posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-02

CONDITIONS: Apnea of Prematurity; Respiratory Distress Syndrome
MeSH Terms: conditions — Apnea; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Discontinue NCPAP after weaning pressures (Active Comparator): After randomization, CPAP pressure will be weaned by 1 every 24hours as long as the subjects continue to meet stability criteria after each wean, until CPAP of 4. If after decrease in CPAP pressure, the subject meets CPAP failure criteria pressure will be increased back to the previous level and after stabilization for 24 hours weaning process will be started again. Once the subject meets stability criteria on CPAP of 4, NCPAP will be stopped and subject will be placed on nasal cannula (NC) according to unit guidelines (max 1 Liter flow, 30% FiO2).
  Interventions: Device: Discontinue NCPAP after weaning pressures
- Discontinue NCPAP without weaning pressures (Active Comparator): After randomization, once the subject meets stability criteria, NCPAP will be stopped and subject will be placed on nasal cannula (NC) according to unit guidelines (max 1 Liter flow, 30% FiO2).
  Interventions: Device: Discontinue NCPAP without weaning pressures

INTERVENTIONS:
Device: Discontinue NCPAP after weaning pressures — After randomization, CPAP pressure will be weaned by 1 every 24hours as long as the subjects continue to meet stability criteria after each wean, until CPAP of 4. If after decrease in CPAP pressure, the subject meets CPAP failure criteria pressure will be increased back to the previous level and after stabilization for 24 hours weaning process will be started again. Once the subject meets stability criteria on CPAP of 4, NCPAP will be stopped and subject will be placed on nasal cannula (NC) according to unit guidelines (max 1 Liter flow, 30% FiO2).
  Arms: Discontinue NCPAP after weaning pressures
Device: Discontinue NCPAP without weaning pressures — After randomization, once the subject meets stability criteria, NCPAP will be stopped and subject will be placed on nasal cannula (NC) according to unit guidelines (max 1 Liter flow, 30% FiO2).
  Arms: Discontinue NCPAP without weaning pressures

SUMMARY:
The purpose of this study is to determine if among infants <30 weeks gestational age on nasal continuous positive airway pressure (NCPAP), whether discontinuing CPAP after gradual reduction in continuous positive airway pressure (CPAP) pressure leads to successful weaning off CPAP when compared to discontinuing CPAP without weaning pressure.

ELIGIBILITY:
Inclusion Criteria:

* All infants < 30 weeks by dates, on NCPAP therapy, on caffeine 10mg/kg daily
* Meet CPAP stability criteria for ≥ 12hours (CPAP 6 cm water (H2O), FiO2 </=0.25 and stable (to maintain sats 85-95%), Respiratory rate consistently less than 60, Mild to no subcostal/intercostal retractions, No Apnea or bradycardia event that requires bag mask ventilation, Less than 3 apnea/brady/desat episodes in any 1 hour period for previous 6 hours, Tolerated time off CPAP during routine CPAP care (~15 min)

Exclusion Criteria:

* Major congenital anomalies including congenital heart disease
* Anomalies that prevent discontinuation of NCPAP
* Undergoing current evaluation for and/or treatment of sepsis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brittany Duyka, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Discontinue NCPAP After Weaning Pressures: After randomization, continuous positive airway pressure (CPAP) will be weaned by 1 every 24 hrs as long as the subjects continue to meet stability criteria after each wean, until CPAP of 4. If after decrease in CPAP pressure the subject meets CPAP failure criteria pressure will be increased back to the previous level and after stabilization for 24 hours weaning process will be started again. Once the subject meets stability criteria on CPAP of 4, NCPAP will be stopped and subject will be placed on nasal cannula (NC) according to unit guidelines (max 1 Liter (1L) flow, 30% FiO2).
- Discontinue NCPAP Without Weaning Pressures: After randomization, once the subject meets stability criteria, NCPAP will be stopped and subject will be placed on nasal cannula (NC) according to unit guidelines (max 1 Liter (1L) flow, 30% FiO2).
Period: Overall Study
Arm/Group | Discontinue NCPAP After Weaning Pressures | Discontinue NCPAP Without Weaning Pressures
Started | 35 | 31
Completed | 29 | 30
Not Completed | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Discontinue NCPAP After Weaning Pressures: After randomization, CPAP pressure will be weaned by 1 every 24 hrs as long as the subjects continue to meet stability criteria after each wean, until CPAP of 4. If after decrease in CPAP pressure, the subject meets CPAP failure criteria (described below) pressure will be increased back to the previous level and after stabilization for 24 hours weaning process will be started again. Once the subject meets stability criteria on CPAP of 4, NCPAP will be stopped and subject will be placed on nasal cannula (NC) according to unit guidelines (max 1L flow, 30% FiO2).
  Discontinue NCPAP after weaning pressures: After randomization, CPAP pressure will be weaned by 1 every 24hours as long as the subjects continue to meet stability criteria after each wean, until CPAP of 4. If after decrease in CPAP pressure, the subject meets CPAP failure criteria (described below) pressure will be increased back to the previous level and after stabilization for 24 hours weaning process will be started again.
- Discontinue NCPAP Without Weaning Pressures: After randomization, once the subject meets stability criteria, NCPAP will be stopped and subject will be placed on nasal cannula (NC) according to unit guidelines (max 1L flow, 30% FiO2).
  Discontinue NCPAP without weaning pressures: After randomization, once the subject meets stability criteria, NCPAP will be stopped and subject will be placed on nasal cannula (NC) according to unit guidelines (max 1L flow, 30% FiO2).
- Total: Total of all reporting groups
Arm/Group | Discontinue NCPAP After Weaning Pressures | Discontinue NCPAP Without Weaning Pressures | Total
Number analyzed (Participants) | 35 | 31 | 66
Age, Continuous [Mean (Full Range); unit: weeks] — corrected gestational age (in weeks) is reported
  weeks | 31.4 [26.1 to 42.4] | 31.1 [27.3 to 35.2] | 31.3 [26.1 to 42.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 15 | 12 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35 | 31 | 66

OUTCOME MEASURES:

1. Primary Outcome: Number of Days on NCPAP or Mechanical Ventilation
Description: Subjects might go on and off NCPAP or mechanical ventilation throughout the 28 days after randomization, and the total number of days will be reported.
Time Frame: from randomization until 28 days post-randomization
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Discontinue NCPAP After Weaning Pressures | Discontinue NCPAP Without Weaning Pressures
Number analyzed (Participants) | 35 | 31
days | 17.3 [14.2 to 20.4] | 12.3 [8.9 to 15.6]

2. Secondary Outcome: Duration of Endotracheal Ventilation
Description: Subjects might go on and off endotracheal ventilation throughout the 28 days after randomization, and the total number of days will be reported.
Time Frame: from randomization until 28 days post-randomization
Population: Data for this measure was not collected.
Arm/Group | Discontinue NCPAP After Weaning Pressures | Discontinue NCPAP Without Weaning Pressures
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants Who Failed to Wean Off NCPAP
Time Frame: from randomization until discharge (about 92 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Discontinue NCPAP After Weaning Pressures | Discontinue NCPAP Without Weaning Pressures
Number analyzed (Participants) | 35 | 31
Participants | 13 | 16

4. Secondary Outcome: Number of Participants Who Developed Bronchopulmonary Dysplasia
Time Frame: from randomization until discharge (about 92 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Discontinue NCPAP After Weaning Pressures | Discontinue NCPAP Without Weaning Pressures
Number analyzed (Participants) | 35 | 31
Participants | 18 | 14

5. Secondary Outcome: Number of Participants Who Developed Necrotizing Enterocolitis
Time Frame: from randomization until discharge (about 92 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Discontinue NCPAP After Weaning Pressures | Discontinue NCPAP Without Weaning Pressures
Number analyzed (Participants) | 35 | 31
Participants | 0 | 0

6. Secondary Outcome: Number of Days of Life at Which Infant Starting Taking All Feeds by Mouth
Time Frame: from randomization until discharge (about 92 days)
Measure: Mean (95% Confidence Interval); unit: number of days of life
Arm/Group | Discontinue NCPAP After Weaning Pressures | Discontinue NCPAP Without Weaning Pressures
Number analyzed (Participants) | 35 | 31
number of days of life | 78 [69 to 88] | 73 [64 to 82]

7. Secondary Outcome: Length of Hospital Stay
Time Frame: from admission to hospital until discharge (about 92 days)
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Discontinue NCPAP After Weaning Pressures | Discontinue NCPAP Without Weaning Pressures
Number analyzed (Participants) | 35 | 31
days | 91.2 [80 to 102.4] | 93.3 [77.8 to 108.7]

8. Secondary Outcome: Number of Participants Who Developed Air Leak Disorders
Description: Air leak disorders include pneumothorax, pneumomediastinum, and pulmonary interstitial emphysema.
Time Frame: from randomization until discharge (about 92 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Discontinue NCPAP After Weaning Pressures | Discontinue NCPAP Without Weaning Pressures
Number analyzed (Participants) | 35 | 31
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: from randomization until discharge (about 92 days)
Description: Only events thought to be related to the intervention are considered to be adverse events.
Arm/Group | Discontinue NCPAP After Weaning Pressures | Discontinue NCPAP Without Weaning Pressures
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/31
Other Adverse Events (participants affected / at risk) | 0/35 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/62/NCT03292562/Prot_SAP_000.pdf